CLINICAL TRIAL: NCT03366649
Title: Improving Mitral Repair for Functional Mitral Regurgitation
Acronym: IMPROVE-FMR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated due to poor enrollment during COVID-19, which also hindered postoperative testing. With insufficient enrollment to meet trial goals, funds were redirected to animal studies on the same clinical issues.
Sponsor: Emory University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Robert Allan Guyton, Professor, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00097939; 1R01HL133667-01A1 (NIH)
Record Dates: First submitted 2017-11-30; First posted 2017-12-08 (Actual); Results first posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2024-12

CONDITIONS: Cardiomyopathy; Cardiovascular Diseases; Congestive Heart Failure; Coronary Artery Disease; Heart Disease; Valvular Heart Disease; Mitral Valve Disease
Keywords: Bypass Surgery; Cardiology; Coronary Artery Bypass Surgery; Mitral Valve Repair; Mitral Valve Surgery; Coronary Revascularization
MeSH Terms: conditions — Cardiomyopathies; Cardiovascular Diseases; Heart Failure; Coronary Artery Disease; Heart Diseases; Heart Valve Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- UMA (Group 1) (Other): Participants in the UMA group will receive an undersizing mitral annuloplasty (UMA).
  Interventions: Procedure: Undersizing Mitral Annuloplasty
- UMA + PMA (Group 2) (Other): Participants in the UMA + PMA group will receive an undersizing mitral annuloplasty (UMA) with papillary muscle approximation (PMA).
  Interventions: Procedure: Undersizing Mitral Annuloplasty; Procedure: Papillary Muscle Approximation
- Retrospectively identified patients (No Intervention): Retrospectively identified patients, who already underwent the standard of care surgery for the lesion of interest at Emory, within 6 months (± 1 month) after the date of their surgery, and are suitable for recruitment to the study for their post-operative research.

INTERVENTIONS:
Procedure: Undersizing Mitral Annuloplasty — Participants will receive a commercially available annuloplasty ring of the surgeon's choice. Sutures are placed around the mitral annulus, and the metallic ring is then implanted onto the mitral annulus to reduce it in size.
  Arms: UMA (Group 1); UMA + PMA (Group 2)
Procedure: Papillary Muscle Approximation — One or two 4-0 pledgeted sutures are used to draw the two papillary muscle tips together to reduce the inter papillary muscle separation (IPMS) before undergoing undersizing mitral annuloplasty.
  Arms: UMA + PMA (Group 2)

SUMMARY:
The investigators are interested in determining the best surgical technique to correct functional mitral regurgitation, as there is currently not one technique that is established to work better than the other.

The technique used in current clinical practice is undersizing mitral annuloplasty (UMA), in which a prosthetic ring is implanted onto the mitral valve to correct the leakage. Though widely adopted, durability of the repair is less, as 58% of the patients present with recurrent FMR within 2 years. There are no specific algorithms to predict who might have UMA failure, but research indicates that some geometric indices might be strong predictors. The investigators are interested in testing the hypothesis that, elevated lateral inter-papillary muscle separation (IPMS) is a predictor of post-UMA recurrence of FMR at 12 months. In the first part of this study, the study team will measure lateral IPMS before surgery and relate to post-surgery FMR severity at discharge/30 days, 6 months and 12 months.

A relatively newer technique is papillary muscle approximation (PMA), in which a suture draws together the two muscles that connect the mitral valve to the heart muscle prior to performing UMA. This reduces the lateral inter-papillary muscle separation (IPMS) and is expected to improve the durability of UMA. In the second part of this study, the investigators will perform PMA and UMA together and determine if FMR severity is reduced at discharge/30 days, 6 months and 12 months.

DETAILED DESCRIPTION:
Functional mitral regurgitation (FMR) is a common heart valve lesion that is observed in patients suffering for cardiomyopathies. Timely surgical repair of FMR can reduce volume overload and potentially improve cardiac function. Durable surgical techniques for FMR repair are lacking. Undersizing mitral annuloplasty (UMA) is the current technique of choice, but its durability is quite poor. Thirty five percent of the repairs fail within one year and 58% fail within 2 years.

One of the probable mechanisms causing UMA failure is elevated lateral inter-papillary muscle separation (IPMS). The study investigators are interested in understanding if the extent of lateral IPMS has a direct impact on the failure rates of UMA at 1 year post surgery. Secondly, the investigators are interested in determining if patients with elevated lateral IPMS benefit from papillary muscle approximation (PMA) along with UMA.

The investigators are interested in determining the best way to correct functional mitral regurgitation, as there is currently not one technique that is established to better than the other. The most common repair technique is called undersizing mitral annuloplasty (UMA), in which a prosthetic ring is implanted onto the mitral valve to correct the leakage. Another more recent technique is papillary muscle approximation (PMA), in which a suture draws together the two muscles that connect the mitral valve to the heart muscle prior to performing UMA. In this research study, the study team is investigating whether they can identify those patients who will benefit from one repair over another.

The primary objective of this protocol is to investigate if pre-operative IPMS is predictive of FMR severity at 12 months after UMA to repair FMR. Furthermore, whether a cut-off value of pre-operative inter-papillary muscle separation can be established to predict patients who might have failure of UMA.

The secondary objective of this protocol is to investigate if adding PMA to UMA is an effective technique in reducing recurrence of FMR at 12 months post-procedure.

ELIGIBILITY:
Inclusion Criteria:

* Mitral regurgitation of moderate or greater severity, as defined by the guidelines of the American Society of Echocardiography (via a transthoracic echo)
* Cardiomyopathy of ischemic or non-ischemic origins, with or without the need for coronary revascularization
* Concomitant right-sided valve repair or replacement (i.e. patients requiring concomitant tricuspid procedures)
* Able to sign informed consent and release of medical information forms

Exclusion Criteria:

* Any evidence of structural (chordal or leaflet) mitral lesions
* Prior mitral valve repair
* Contraindication for cardiopulmonary bypass
* Clinical signs of cardiogenic shock at the time of randomization
* ST-segment elevation myocardial infarction within 14 days before inclusion in this study
* Congenital heart disease, except patent foramen ovale (PFO) or atrial septal defect (ASD)
* Chronic renal insufficiency defined by creatinine ≥ 3.0 or chronic renal replacement therapy, who are contraindicated for cardiac surgery
* Recent history of psychiatric disease that is likely to impair compliance with the study protocol, in the judgement of the investigator
* Pregnancy at the time of randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Guyton, MD, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Emory St. Joseph's Hospital, Atlanta, Georgia

REFERENCES:
- [Background] Kalra K, Wang Q, McIver BV, Shi W, Guyton RA, Sun W, Sarin EL, Thourani VH, Padala M. Temporal changes in interpapillary muscle dynamics as an active indicator of mitral valve and left ventricular interaction in ischemic mitral regurgitation. J Am Coll Cardiol. 2014 Nov 4;64(18):1867-79. doi: 10.1016/j.jacc.2014.07.988. Epub 2014 Oct 27. PMID 25444139
- [Background] Michler RE, Smith PK, Parides MK, Ailawadi G, Thourani V, Moskowitz AJ, Acker MA, Hung JW, Chang HL, Perrault LP, Gillinov AM, Argenziano M, Bagiella E, Overbey JR, Moquete EG, Gupta LN, Miller MA, Taddei-Peters WC, Jeffries N, Weisel RD, Rose EA, Gammie JS, DeRose JJ Jr, Puskas JD, Dagenais F, Burks SG, El-Hamamsy I, Milano CA, Atluri P, Voisine P, O'Gara PT, Gelijns AC; CTSN. Two-Year Outcomes of Surgical Treatment of Moderate Ischemic Mitral Regurgitation. N Engl J Med. 2016 May 19;374(20):1932-41. doi: 10.1056/NEJMoa1602003. Epub 2016 Apr 3. PMID 27040451
- [Background] Kron IL, Hung J, Overbey JR, Bouchard D, Gelijns AC, Moskowitz AJ, Voisine P, O'Gara PT, Argenziano M, Michler RE, Gillinov M, Puskas JD, Gammie JS, Mack MJ, Smith PK, Sai-Sudhakar C, Gardner TJ, Ailawadi G, Zeng X, O'Sullivan K, Parides MK, Swayze R, Thourani V, Rose EA, Perrault LP, Acker MA; CTSN Investigators. Predicting recurrent mitral regurgitation after mitral valve repair for severe ischemic mitral regurgitation. J Thorac Cardiovasc Surg. 2015 Mar;149(3):752-61.e1. doi: 10.1016/j.jtcvs.2014.10.120. Epub 2014 Nov 6. PMID 25500293
- [Background] Acker MA, Parides MK, Perrault LP, Moskowitz AJ, Gelijns AC, Voisine P, Smith PK, Hung JW, Blackstone EH, Puskas JD, Argenziano M, Gammie JS, Mack M, Ascheim DD, Bagiella E, Moquete EG, Ferguson TB, Horvath KA, Geller NL, Miller MA, Woo YJ, D'Alessandro DA, Ailawadi G, Dagenais F, Gardner TJ, O'Gara PT, Michler RE, Kron IL; CTSN. Mitral-valve repair versus replacement for severe ischemic mitral regurgitation. N Engl J Med. 2014 Jan 2;370(1):23-32. doi: 10.1056/NEJMoa1312808. Epub 2013 Nov 18. PMID 24245543

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Efforts were made to include post-surgery patients and those from prior years. However, required preoperative imaging was unavailable, preventing preop vs. follow-up comparisons. No participants were enrolled in UMA + PMA (Group 2), and no retrospectively identified patients were included in Group 3.
Groups:
- No Intervention: Retrospectively Identified Patients: Retrospectively identified patients, who already underwent the standard of care surgery for the lesion of interest at Emory, within 6 months (± 1 month) after their surgery, and suitable for recruitment to the study for their post-operative research.
Period: Overall Study
Arm/Group | UMA (Group 1) | UMA + PMA (Group 2) | No Intervention: Retrospectively Identified Patients
Started | 34 | 0 | 0
Completed | 26 | 0 | 0
Not Completed | 8 | 0 | 0
Not completed — Failed preoperative screening | 4 | 0 | 0
Not completed — Had concomitant valves replacements, therefore not included in data analysis | 4 | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | UMA (Group 1)
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.6 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 16
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Change in FMR Severity
Description: The Severity (grade 0 to 4+) of mitral regurgitation of mitral regurgitation is measured using cardiac echocardiography and/or MRI (per physician's discretion).
  Grade 0: None Grade 1 (Mild): Small, restricted jet of regurgitation with minimal impact on the heart's function. Typically, no symptoms and normal or near-normal left ventricular function.
  Grade 2 (Moderate): Moderate jet size with some effect on the heart, but symptoms may still be absent or minimal. Mild to moderate left ventricular dilation may be present.
  Grade 3 (Moderately Severe): Larger jet, more significant regurgitation, potentially causing mild heart failure symptoms or moderate dilation of the left ventricle.
  Grade 4 (Severe): A large, prominent jet of regurgitation that significantly impacts heart function, often resulting in severe symptoms and marked left ventricular dilation.
Time Frame: Pre-Intervention and Post-Intervention (12 Months)
Population: Data is available only for the 12-month follow-up, as other data was unavailable due to many follow-ups occurring during the COVID pandemic.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | UMA (Group 1)
Number analyzed (Participants) | 26
score on a scale
  Baseline | 2.7 (0.8)
  12 months post-intervention | 0.7 (0.7)

2. Secondary Outcome: Mortality Rate
Description: The number of participants who are deceased will be collected throughout the study at discharge and planned follow up visits.
Time Frame: Post-Intervention (Up to 20 Days), Post-Intervention (Month 6), Post-Intervention (Month 12)
Measure: Count of Participants; unit: Participants
Arm/Group | UMA (Group 1)
Number analyzed (Participants) | 26
Participants
  up to 20 days post-Intervention | 0
  12 months post-intervention | 0

3. Secondary Outcome: Number of Major Adverse Cardiac Events (MACE)
Description: MACE is defined as a composite of clinical events comprised of the following:
  * Death
  * Stroke
  * Worsening heart failure (+1 New York Heart Association (NYHA) class)
  * Congestive heart failure (CHF) hospitalization
  * Mitral valve re-intervention
Time Frame: Up to 12 months post -intervention
Population: Participants with valid data.
Measure: Count of Participants; unit: Participants
Arm/Group | UMA (Group 1)
Number analyzed (Participants) | 26
Participants
  Congestive heart failure (CHF) hospitalization | 1
  Death | 0
  Mitral valve re-intervention | 0
  Stroke | 0
  Worsening heart failure (+1 New York Heart Association (NYHA) class): number analyzed (Participants) | 19
  Worsening heart failure (+1 New York Heart Association (NYHA) class) | 0

4. Secondary Outcome: Change in Quality-of-Life Scale Score
Description: Participants will be asked to measure their perceived quality of life on a scale from 0 to 100 where 0 indicates "worst imaginable health state" and 100 indicates "best imaginable health state".
Time Frame: Baseline, Post-Intervention (Month 6), Post-Intervention (Month 12)
Population: Participants who completed the questionnaires within the specific study window. Data is available only for the 12-month follow-up, as other data was unavailable due to many follow-ups occurring during the COVID pandemic.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | UMA (Group 1)
Number analyzed (Participants) | 10
Score on a scale
  Baseline | 69.0 (19.0)
  Post-Intervention (Month 12): number analyzed (Participants) | 8
  Post-Intervention (Month 12) | 76.9 (16.9)

5. Secondary Outcome: Change in Minnesota Living With Heart Failure (MLHF) Questionnaire Score
Description: The Minnesota Living with Heart Failure Questionnaire is a 21-item questionnaire that asks participants to describe how much their heart failure has affected life during the past month (4 weeks). Participants are asked if their heart failure prevented them from living as they want when completing daily tasks. Responses are rated on a scale from 0 to 5; 0 represents "no", 1 represents "very little" and 5 represents "very much" on a continuum. The MLHF score is obtained by summing the subjects responses. A minimum score is 0 indicating no affect to life and a maximum score is 105 indicating the greatest affect to life.
Time Frame: Baseline, Post-Intervention (Month 12)
Population: Participants who answered the specific questionnaires within the specific study window. Data is available only for the 12-month follow-up, as other data was unavailable due to many follow-ups occurring during the COVID pandemic.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | UMA (Group 1)
Number analyzed (Participants) | 11
score on a scale
  Baseline | 44.2 (31.3)
  12 months Post-Intervention | 30.9 (28.0)

6. Secondary Outcome: Change in Functional Status Assessed by 6-Minute Walk Test (6MWT)
Description: Functional status will be measured by a 6-minute walk test, which assesses the distance walked (in feet) on a flat, hard surface in a period of 6 minutes (the 6MWD). The test is used for preoperative and postoperative evaluation and for measuring the response to therapeutic interventions for pulmonary and cardiac disease. Optimal reference equations from healthy population-based samples using standardized 6MWT methods are not yet available. A low 6MWD is nonspecific and nondiagnostic. When the 6MWD is reduced, a thorough search for the cause of the impairment is warranted.
Time Frame: Baseline, Post-intervention (Month 6), Post-Intervention (Month 12)
Population: Participants who completed the study procedure. Data is available only for the 12-month follow-up, as other data was unavailable due to many follow-ups occurring during the COVID pandemic.
Measure: Mean (Standard Deviation); unit: feet
Arm/Group | UMA (Group 1)
Number analyzed (Participants) | 11
feet
  Baseline: number analyzed (Participants) | 6
  Baseline | 1048.4 (293.7)
  12 months Post-Intervention | 1210.6 (203.6)

7. Secondary Outcome: All Cause Readmission Rate
Description: Readmission rate will be calculated for any cause within the first 30 days following surgery throughout the duration of the study.
Time Frame: Post Surgery (Up to 30 Days)
Population: Participants with valid data.
Measure: Count of Participants; unit: Participants
Arm/Group | UMA (Group 1)
Number analyzed (Participants) | 26
Participants
  Post-Surgery (up to 30 days) | 2
  Post-Surgery (30 days through 12 Months) | 4

8. Secondary Outcome: Heart Failure Readmission Rate
Description: Readmission rate will be calculated for heart failure after 30 days following surgery throughout the duration of the study. Classification of readmission as heart failure related requires at least 2 out of the following signs and symptoms of acute decompensated heart failure:
  * Dyspnea felt related to HF
  * Treatment with intravenous diuretic, vasodilator or inotropic therapy
  * X ray evidence of pulmonary edema or pulmonary vascular congestion
  * Rales on physical exam
  * Pulmonary capillary wedge pressure (PCWP) or LVEDP > 18mm Hg
Time Frame: Post Surgery (Up to 30 Days)
Population: Participants with valid data.
Measure: Count of Participants; unit: Participants
Arm/Group | UMA (Group 1)
Number analyzed (Participants) | 26
Participants | 0

9. Secondary Outcome: Change in Left Ventricular Volume
Description: Change in left ventricular volume at 6- and 12-month post-intervention compared to baseline as measured by as measured by the left ventricular end-diastolic diameter determined by echocardiogram.
Time Frame: Baseline, Post-Intervention (Month 6), Post-Intervention (Month 12)
Population: Participants with valid data. Data is available only for the 12-month follow-up, as other data was sparse due to many follow-ups occurring during the COVID pandemic.
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | UMA (Group 1)
Number analyzed (Participants) | 26
centimeters
  Baseline | 5.4 (0.8)
  12 months Post-Intervention | 4.8 (0.8)

10. Secondary Outcome: Change in Ejection Fraction
Description: Change in left ventricular ejection fraction at 12- months post-intervention compared to baseline as measured by echocardiogram.
Time Frame: Baseline, Post-Intervention (Month 12)
Population: Participants who had adequate echocardiograms to complete this evaluation.
Measure: Mean (Standard Deviation); unit: percentage of ejection fraction
Arm/Group | UMA (Group 1)
Number analyzed (Participants) | 26
percentage of ejection fraction
  Baseline | 45 (14)
  12 months post-intervention | 46 (14)

11. Secondary Outcome: Change in Left Ventricular Mass
Description: Change in left ventricular mass at 12 months post intervention compared to baseline as measured by cardiac MRI.
Time Frame: Baseline, Post-Intervention (Month 12)
Population: Some MRIs were performed but not analyzed, as these were research trial MRIs. The original PI and a research post-doc who were the expert analysts, left before reading the MRIs. Only eight patients had both pre- and post-MRIs. Outsourcing analysis was too costly, and meaningful comparisons weren't possible with such a small sample, so the MRIs were not read for the study.
Arm/Group | UMA (Group 1)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Considering the observational nature of this study, and the absence of any experimental procedures, adverse event (AE) reporting was limited only to those events that occurred from the specific non-standard-of-care lab procedures that were performed at 6- and 12-month visits.
Description: An adverse event (AE) is any undesirable clinical occurrence related to a non-standard-of-care study intervention. Pre-existing or associated Conditions with standard care are not AEs unless they change in nature, severity, or degree. AEs are typically reported in trials involving experimental interventions. In this observational study, AE reporting was limited to events from non-standard-of-care lab procedures at the 6- and 12-month visits, none of which were related to those procedures.
Arm/Group | UMA (Group 1)
All-Cause Mortality (participants affected / at risk) | 0/26
Serious Adverse Events (participants affected / at risk) | 4/26
Other Adverse Events (participants affected / at risk) | 0/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | UMA (Group 1) (N=26)
Atrial fibrillation + congestive heart failure (CHF) (Cardiac disorders) | 1 (1) — Hospital admission due to Atrial fibrillation + congestive heart failure (CHF)
Atrial Flutter (Cardiac disorders) | 1 (1) — Hospital admission due to Atrial Flutter
Acute cholecystitis with perforated gallbladder (Gastrointestinal disorders) | 1 (1) — Hospital admission due to acute cholecystitis with perforated gallbladder
Syncope (General disorders) | 1 (1) — Hospital admission due to syncope.

LIMITATIONS AND CAVEATS:
Funds were granted for a clinical study led by the original PI, but enrollment halted during the pandemic. Follow-up was difficult, preventing study procedures, and preoperative imaging was lacking, preventing comparisons. The PI left in April 2023, leaving no expert MRI analysts for limited data. Dr. Guyton took over 8 months before the study was terminated. The NIH redirected funding to large animal studies and computational analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-06-17): https://cdn.clinicaltrials.gov/large-docs/49/NCT03366649/Prot_SAP_001.pdf
  • Informed Consent Form (2023-02-20): https://cdn.clinicaltrials.gov/large-docs/49/NCT03366649/ICF_002.pdf